CLINICAL TRIAL: NCT00205621
Title: Positron Emission Tomography of Cerebral Amyloid Load as a Potential Diagnostic Marker for Pre-Symptomatic Alzheimer's Disease.
Brief Title: Positron Emission Tomography of Amyloid in Alzheimer's Disease
Status: Suspended | Phase: Phase 1 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2005/90
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2005-08

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; amyloid; PET; PIB; FDDNP
MeSH Terms: conditions — Alzheimer Disease | interventions — Positron-Emission Tomography

INTERVENTIONS:
Device: Positron Emission Tomography

SUMMARY:
In this study in-vivo quantification of amyloid load will be performed in patients with AD, MCI and normal controls with Positron Emission Tomography. For this the PET tracers [11C]PIB and [18F]FDDNP will be compared.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a fatal neurodegenerative disorder characterized by progressive impairment in daily life, cognitive deterioration, and a variety of neuropsychiatric and behavioural symptoms. The diagnosis of AD is based on clinical criteria, but these have low sensitivity and specificity for AD in the early stages of the disease. Therefore, there is a great need for a method to identify the pathological process of AD at an earlier, preclinical stage. In-vivo imaging and quantification of pathological beta-amyloid (Aß) accumulation may provide such a method as the production and accumulation of Aß is thought to be central to the pathogenesis of AD. The view is widely held that Aß may be present in the brain at sublethal concentrations for extended periods before the overt manifestation of AD. Therefore, early, in-vivo detection of pathological Aß accumulation is warranted and may identify subjects at risk for AD. Neuroimaging with Positron Emission Tomography (PET) permits in-vivo imaging and quantification of cerebral amyloid load, which is a novel application of PET. Recently, several PET tracers ([18F]FDDNP and [11C]PIB) have been developed for this purpose and the first clinical studies in patients with AD are encouraging. For both tracers, many methodological issues still need to be resolved and the clinical value of in-vivo amyloid imaging remains to be established. The most important objectives of this project are twofold: to provide an independent and unbiased evaluation of the value of in-vivo amyloid imaging in the (early) diagnosis of AD and to optimize methods for quantification of the in-vivo cerebral amyloid load. To investigate the value in the early diagnosis, identification of subjects at risk for AD is essential. Patients with amnestic mild cognitive impairment (MCI), i.e patients suffering only from memory problems but without the other symptoms of AD, are recruited for this purpose. MCI is a disease state considered to be a transitional state between normal aging and dementia. It is generally accepted that the ability to identify the presence of Alzheimer type pathology in the MCI stage will benefit disease management. Twenty patients with amnestic MCI, 15 patients with AD and 15 age and sex matched healthy controls will be included in this study. Only consecutive new patients fulfilling criteria of amnestic MCI will be included. Patients with MCI will remain under clinical observation during two years after participation in order to monitor conversion to clinical dementia. All subjects will receive [11C]PIB and [18F]FDDNP PET scans on a single day. In addition, patients will receive a [18F]FDG PET scan. Furthermore, an MRI scan, a neuropsychological evaluation and CSF analysis for diagnostic purposes will be performed in all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of probable Alzheimer's disease (NINCDS-ADRDA criteria)
* Clinical diagnosis of MCI according to the criteria of Petersen
* Age between 60 and 80 years
* Written informed consent of each subject.
* Hb must be >8 mmol \ litre at the time of the screening for males and >7 mmol\litre for females.
* Weight >50 kg
* All subjects have to be "wilsbekwaam"

Exclusion Criteria:

* Any clinical significant abnormality of any clinical laboratory test
* Any subject who has received any investigational medication within 30 days prior to the start of this study, or who is scheduled to receive an investigational drug.
* Major psychiatric or neurological disorder other than AD
* History of AD in first degree relatives (controls only)
* History of alcohol and/or drug abuse (DSM-IV criteria)
* Any sign of cardiovascular disease including ECG
* Claustrophobia
* Mini Mental State Score below 20
* Use of non-steroid anti-inflammatory drugs
* Abnormalities on MRI other than white matter changes or an incidental small lacunar lesion.
* Blood donation within 3 months before the scan day
* Metal objects in or around the body (braces, pacemaker, metal fragments)
* Use of antithrombotics and ASA
* Fall ≤ 6 months or any relevant gait disorder
* Need for elective surgery ≤ 3 months

Ages: 60 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-10; Study Completion 2009-12

PRIMARY OUTCOMES:
quantification of amyloid binding

CONTACTS AND LOCATIONS:
Overall Officials: Bart van Berckel, MD; PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands